CLINICAL TRIAL: NCT00905411
Title: Pacific Kids DASH for Health
Acronym: PacDASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 2008-55215-18821; 2007-04557
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2011-11

CONDITIONS: Overweight; Blood Pressure
Keywords: Overweight; blood pressure; DASH diet; Pacific; children
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Control / Usual Care (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: PacDASH intervention

INTERVENTIONS:
Behavioral: PacDASH intervention — Effect of the PacDASH intervention on nutrition and physical activity behavior of children.
  15 months study.
  Arms: Intervention

SUMMARY:
The increasing prevalence of childhood overweight has been found to be related to decreased levels of physical activity (PA) and increased energy content of the diet. Childhood offers an opportunity to develop and support health-promoting behaviors. Pacific Kids DASH for Health (PacDASH) is a community-based intervention that links food, PA, and health, and targets overweight children in Hawaii with a goal of preventing further weight gain. Components of the intervention include a food and PA prescription delivered by physicians at community-based health centers complemented with a toolbox of activities, behaviorally tailored messages, and PacDASH educational materials. This project will extend and apply the nationally recommended DASH eating pattern to children and the growing population of Asians and Pacific Islanders. The investigators will incorporate culturally preferred foods, recipes, and PA messages that meet DASH and other national guidelines. The approach will target child food behaviors and social and environmental cues that are important to making healthy food and PA choices and will provide steps to behavior change. Farmers markets at participating health centers are a support resource for activities. Providing access to, coupons for, and guidance about selecting and preparing fresh fruits and vegetables at a convenient health center farmers market will support increased intake of nutrient-rich foods among these children who are overweight and at risk for obesity.

Pacific Islanders are among the world's most obese populations while Asians, although of relatively low body mass index (BMI), carry much of their body fat in the upper body and exhibit greater health risk at the same BMI. Through this project, the investigators hope to learn more about body size and composition in children of the Pacific Region for whom there are few national data. In addition, evaluate the effectiveness of a community-based intervention within a health care system on managing overweight in children.

DETAILED DESCRIPTION:
INTRODUCTION The ethnic groups of the Pacific Region are predominantly Pacific Islander and Asian.

Pacific Islanders (PacIsl) are among the world's most obese populations while Asians, although of relatively low body mass index (BMI), carry much of their body fat in the upper body and exhibit greater health risk at the same BMI. Childhood offers an opportunity to develop and support health-promoting behaviors. This project will extend and apply the nationally recommended DASH eating pattern 115, developed for White, African American and Hispanic adults, to children and to the growing population of Asians and PacIsl. We will incorporate culturally-preferred foods, recipes, and physical activities that meet DASH and other national guidelines, with adaptations for children. We will develop the Pacific Kids DASH for Health (PacDASH) intervention in Hawaii, where the majority is of Asian and PacIsl ancestry.

Linking food and health systems is critical to prevent obesity. The PacDASH intervention will include a food and physical activity (PA) prescription delivered by a physician at a community-based health center (HC), in partnership with farmers' markets (FM) that are based at the HC, and complemented with a toolbox of related activities. The intervention approach supports child food behaviors and social and environmental cues, which are important to making healthy food and PA choices. Linking physicians and health with farmers and food at a convenient HC FM will support increased intake of nutrient-rich, less energy dense foods among children of understudied ethnic groups who are at high risk for obesity.

Project Goal Our goal is to develop and evaluate the effectiveness of a community-based intervention that links food and health, and targets children of the Pacific Region who are overweight, in order to slow and prevent further weight gain (for children to "grow into their weight").

Specific Objectives

1. To develop and evaluate the impact of the PacDASH intervention on preventing weight gain and improving blood pressure in children of the Pacific Region.

   1. To further develop and test the Pacific Tracker (PacTrac) dietary assessment and education tool by incorporating updated MyPyramid 112 reference data and educational output, and
   2. To enhance PacTrac with an expert system (ES) of behaviorally-tailored messages and output.
   3. To evaluate the effect of the PacDASH intervention on nutrition and physical activity behavior of children.
2. To describe environmental, social, economic and cultural factors associated with body size and composition of children of the Pacific Region, for whom there are few national data.

   1. To examine body size and composition of children of the Pacific Region according to several measures.
   2. To examine the influence of individual PacIsl ethnic groups on body size and composition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 - 8 years old
2. >85th up to 98th BMI-for-age percentile (overweight)
3. Children with a primary care provider at MAP
4. Lives on Oahu
5. Due for, or scheduled for, a well-child/physical exam visit during months of the pilot study

Exclusion Criteria:

1. Diabetes Mellitis
2. Polycystic Ovarian Syndrome
3. Gastroesophageal Reflux
4. Gallbladder disease
5. Non alcoholic fatty liver disease
6. Pseudo Tumor cerebri
7. Slipped capital femoral epiphysis
8. Blount's disease
9. Obstructive Sleep Apnea/Sleep Disturbance
10. Other chronic disease conditions that would affect participation

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Develop/evaluate effectiveness of a community-based intervention targets children of the Pacific Region who are overweight in order to slow and prevent further weight gain (for children to "grow into their weight") | Feb 2008 - Feb 2012

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Novotny, PhD,RD, Principal Investigator — Kaiser Permanente Center for Health Research Hawaii, University of Hawaii, Human Nutrition, Food, Animal Sciences Department
Locations (1):
- Kaiser Permanente Center for Health Research, Hawaii, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Novotny R, Nigg CR, Li F, Wilkens LR. Pacific kids DASH for health (PacDASH) randomized, controlled trial with DASH eating plan plus physical activity improves fruit and vegetable intake and diastolic blood pressure in children. Child Obes. 2015 Apr;11(2):177-86. doi: 10.1089/chi.2014.0141. Epub 2015 Feb 11. PMID 25671796